CLINICAL TRIAL: NCT00003757
Title: Rituximab (IDEC-C2B8, Mabthera) in Patients With Hairy Cell Leukemia Relapsing After Treatment With 2-Chlorodeoxyadenosine (CDA)
Brief Title: Rituximab in Treating Patients With Refractory or Recurrent Hairy Cell Leukemia Following Cladribine Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: SAKK 31/98; SWS-SAKK-31/98; EU-98073
Record Dates: First submitted 1999-11-01; First posted 2003-04-30 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Leukemia
Keywords: progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Hairy Cell | interventions — Rituximab

INTERVENTIONS:
Biological: rituximab

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of monoclonal antibody therapy consisting of rituximab in treating patients with refractory or recurrent hairy cell leukemia following cladribine therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the rate of complete and partial remission, remission duration, and relapse free survival after treatment with rituximab in patients with refractory or recurrent hairy cell leukemia who previously received cladribine.
* Determine the acute and long term toxicity of rituximab in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive rituximab IV over several hours once a week for 4 weeks.

Patients are followed every 3 months for 3 years and every 6 months thereafter.

PROJECTED ACCRUAL: A total of 8-25 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven hairy cell leukemia (HCL)

  * Classic HCL

    * Hairy cells in the bone marrow and/or peripheral blood which co-express CD20/CD25 or CD20/CD11c, and/or which are positive for tartrate resistant acid phophatase (TRAP)
  * Prolymphocytic HCL variant

    * Lymphoid cells in the bone marrow and/or peripheral blood with morphology intermediate between typical hairy cells and prolymphocytes, which co-express CD20/CD11c but lack CD25 expression, and which are negative for TRAP
* Progressive or recurrent disease after prior treatment with cladribine

  * Greater than 1 month since standard dose cladribine OR
  * Greater than 3 months since low dose cladribine

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2.0 mg/dL

Renal:

* Creatinine no greater than 2.3 mg/dL

Cardiovascular:

* No serious cardiac disease

Other:

* No acute or chronic infection
* HIV negative
* No psychosis
* Not pregnant or nursing
* No other prior or concurrent malignancy except carcinoma in situ of the cervix or basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* Recovered from prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* Recovered from prior therapy
* No concurrent cytoreductive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1998-02; Primary Completion 2002-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert von Rohr, MD, Study Chair — Klinik Hirslanden, Zurich
Locations (1):
- Klinik Hirslanden, Zurich, Switzerland

REFERENCES:
- [Result] Zenhausern R, Simcock M, Gratwohl A, Hess U, Bargetzi M, Tobler A; Swiss Group for Clinical Cancer Research (SAKK). Rituximab in patients with hairy cell leukemia relapsing after treatment with 2-chlorodeoxyadenosine (SAKK 31/98). Haematologica. 2008 Sep;93(9):1426-8. doi: 10.3324/haematol.11564. Epub 2008 Jul 4. No abstract available. PMID 18603561